CLINICAL TRIAL: NCT04471311
Title: Safety and Efficacy of Prophylactic Resorbable Biosynthetic Mesh Following Midline Laparotomy in Clean/Contaminated Field: Protocol for a Multicenter Randomized Double Blind Prospected Trial.
Brief Title: Safety and Efficacy of Prophylactic Re-sorbable Biosynthetic Mesh Following Midline Laparotomy in Clean/Contaminated Field.
Acronym: Parthenope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Head of Bariatric Unit, Azienda Sanitaria Locale Napoli 2 Nord
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1872020
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Incisional Hernia After Midline Laparotomy
Keywords: Incisional Hernia; Midline laparotomy; Contaminated wound
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Intervention Model Description: THIS IS A CONTROLLED RANDOMIZED STUDY OF BINARY SUPERIORITY OUTCOME IN PARALLEL GROUPS. 302 PATIENTS ARE REQUIRED TO HAVE A 95% CHANCE OF DETECTING, AS SIGNIFICANT AT THE 5% LEVEL, A DECREASE IN THE PRIMARY OUTCOME MEASURE FROM 18% (INCISIONAL HERNIA RATE) IN THE CONTROL GROUP TO 5%(INCISIONAL HERNIA RATE) IN THE EXPERIMENTAL GROUP.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary closure of midline laparotomy (No Intervention): Primary closure of midline laparotomy
- Sub-lay mesh supported closure (Experimental): Sub-lay permanent mesh supported the closure
  Interventions: Procedure: Sub-lay mesh supported closure; Device: BIO-A (GORE) mesh

INTERVENTIONS:
Procedure: Sub-lay mesh supported closure — A 4 cm space is created between posterior rectus sheath and rectus muscle, widening 2 cm at each side of midline. Both posterior rectus sheath edges are sutured using a running slowly absorbable suture. Above the arcuate line, posterior layer is reinforced suturing the peritoneum and the posterior rectus sheath; below the arcuate line, the posterior layer is reinforced suturing the peritoneum and the trasversalis fascia. Anterior layer is re-established suturing the anterior rectus sheath. A 3 cm BIO-A Mesh strip is sutureless placed between the posterior rectus sheath and the rectus muscle with an overlap of 1,5 cm at each side. In laparotomies >20 cm two stripes of 15 cm each is designed. The midline anterior rectus sheath is closed using a running slowly absorbable suture , covering the mesh.
  Arms: Sub-lay mesh supported closure
Device: BIO-A (GORE) mesh — 3 cm BIO-A Mesh strip
  Arms: Sub-lay mesh supported closure

SUMMARY:
The aim of the present study is to analyse the feasibility, safety and IH rate using a prophylactic sublay biosynthetic BIO-A (GORE) mesh in order to prevent incisional hernia following midline laparotomy in clean-contaminated and contaminated wounds. The study was designed as a double-blind randomized controlled trial comparing the running suture alone to the running suture reinforced with biosynthetic mesh (BIOA) in sub lay position.

DETAILED DESCRIPTION:
Incisional Hernia (IH) is one of the most frequent postoperative complications in abdominal surgery causing significant morbidity and even mortality. The risk of developing an IH following primary elective midline laparotomy is reported to be between 5 and 20 percent. Risk factors for developing IH are both patient and surgery related. Patient factors include diabetes, smoking, obesity, chronic corticosteroids use and connective tissue disorders, comprised the presence of an Abdominal Aortic Aneurysm (AAA). Surgery related factors include type of laparotomy, type of surgery, wounds classification, suture material used to close the laparotomy and the suture length to wound length ratio (SL/WL).

In patients carrying AAA and/or obesity and/or contaminated wounds, incidence rises to 39% (6,7). Besides the negative impact of incisional hernia regarding the patients' quality of life, the direct costs of hernia repair and indirect cost of IH (sick leave) are an important burden for the health care system.

Several groups investigated the role of prophylactic mesh placement in the prevention of IH occurrence. A positive conclusion was reached by two systemic reviews. On the other side, surgeons are mostly reluctant to implant permanent material in patients undergoing a contaminated ventral hernia repair for the increased risk of postoperative infections, bowel adhesions, mesh extrusion and/or erosion, fistula formation, seroma development and pain.

Recently, a retrospective study by Carbonell et al. investigated the feasibility and outcomes of open ventral hernia repairs performed with a polypropylene mesh in the retro-rectus position in clean-contaminated and contaminated fields, reporting a 30-day surgical site infection rate of 7.1 and 19.0% respectively. The most appropriate mesh for hernia repair in clean-contaminated and contaminated fields is not as clear .

Some other authors proposed the implant of Biological Meshes (BM) in contaminated and dirty wounds, but their high costs limited their use. Moreover, data about long-term durability of biologic grafts used in case of complex abdominal wall reconstruction are not clearly defined. The so-called biosynthetic meshes (BSM) may, actually, offer advantages when challenging with bacterial colonization during complex abdominal wall reconstruction.

The GORE BIO-A Tissue Reinforcement is a BSM composed of a bio-absorbable polyglycolide-trimethylene carbonate copolymer, which is gradually absorbed by the body.

The aim of the present study is to analyse the feasibility, safety and IH rate using a prophylactic sublay biosynthetic BIO-A (GORE) mesh in order to prevent incisional hernia following midline laparotomy in clean-contaminated and contaminated wounds. The study was designed as a double-blind randomized controlled trial comparing the running suture alone to the running suture reinforced with biosynthetic mesh (BIOA) in sub lay position.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Clean-contaminated, contaminated wounds • midline laparotomy >10 cm
* Informed consent

Exclusion Criteria:

* age < 18 years;
* life expectancy < 24 months (as estimated by the operating surgeon), - • pregnancy
* immunosuppressant therapy within 2 weeks before surgery
* clean and dirty wounds
* wound length<10 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Incisional Hernia at Ultrasound examination | 3 months
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | 6 months
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | 12 months
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | 24 months
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Clinical examination | 3 months
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | 6 months
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | 12 months
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | 24 months
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar

SECONDARY OUTCOMES:
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pizza, Study Director — Azienda Sanitaria Locale Napoli 2 Nord
Locations (1):
- francesco Pizza, Naples, Italy

IPD SHARING:
Plan to Share IPD: No